CLINICAL TRIAL: NCT00401414
Title: CReating an Optimal Warfarin Nomogram (CROWN) Trial
Brief Title: Study to Develop a Reliable Nomogram That Incorporates Clinical and Genetic Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Newton-Wellesley Hospital (Other); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Mark Alan Creager, MD, Director, Vascular Center, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-001896
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-07

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis; Atrial Fibrillation
Keywords: Warfarin; Thrombosis; Genetics; Nomogram; Pulmonary Embolism; Deep Vein Thrombosis; Dosing; INR; Anticoagulation; Therapy; Orthopedic Surgery
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Atrial Fibrillation; Thrombosis | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Warfarin (Experimental): We will develop a nomogram for warfarin dosing that uses rapid turnaround genetic testing and monthly nomogram modification (if necessary) to achieve effective and safe warfarin induction and maintenance. More than 70% of the time, we will maintain warfarin naïve patients within the target therapeutic range. The percent of time in the therapeutic range will be analyzed beginning 2 weeks after initiation of warfarin. Analyses will be stratified by the indication for anticoagulation.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — 2 mg tablets take as directed by study staff (based on INR)

SUMMARY:
In this research study, the investigators are trying to find a better way to set the dose of a common blood-thinning medication.

Patients with blood clots or a risk of blood clots (or stroke) sometimes have to take an approved medication called warfarin. Warfarin is a commonly prescribed, approved blood thinning medicine taken by mouth. There is a certain level of warfarin that is best for each patient at a particular time. It is hard for a doctor to choose and maintain the right dose of warfarin for each patient. Too much or too little warfarin in the blood can cause serious health problems.

A "nomogram" is a tool that helps doctors decide on the right dose of warfarin. The usual way for finding the right dose of warfarin is for doctors to take an educated guess and use a "trial and error" approach. Patients have frequent blood tests to help doctors keep track of how well the dose level is working.

Up until now, if a patient had good blood test results over half of the time, that was as well as doctors could do. The purpose of this study is to see whether the investigators can create a reliable new warfarin nomogram that will allow them to dose a patient correctly more often, perhaps about 3 times out of 4. The nomogram the investigators are studying uses information about a patient's health and genes to decide on the best dose of warfarin.

The investigators don't yet have a reliable, safe way to choose the correct dose. In this study, the investigators will use a genetic blood test to try to find a better way. Genes are the parts of each living cell that allow characteristics to be passed on from parents to children. The investigators know that people with certain genes seem to respond to warfarin in a certain way. From a blood sample, the investigators can look at patients' genes and try to predict the response to the blood-thinning medication.

There will be about 500 subjects taking part in this study. They will come from participating Partners' Hospitals, including Brigham and Women's Hospital, Massachusetts General Hospital, Faulkner Hospital, Newton-Wellesley Hospital, Spaulding Rehabilitation Hospital, and North Shore Medical Center. The U.S. Food and Drug Administration (FDA) has approved warfarin for use as a blood thinner.

DETAILED DESCRIPTION:
This is Phase 1 of a 3-phase plan in which we will ultimately test whether rapid turnaround genetic testing can improve the safety and efficacy of warfarin anticoagulation in warfarin naïve patients who are being newly induced and maintained on warfarin. Each of the phases will address a specific and progressively more ambitious question.

Phase 1 will be a 500-patient cohort study to determine whether we can develop a reliable nomogram that incorporates clinical and genetic information to maintain patients within the target therapeutic range more often than 70% of the time, the conventional historical benchmark for excellence in warfarin dosing.

BACKGROUND:

Warfarin was patented in 1948 and was introduced commercially in 1954. In 2004, more than 24 million prescriptions were written for warfarin in the United States alone. Warfarin constitutes the 20th most frequently prescribed drug in the United States. This is remarkable, because few drugs have had a life cycle as long as warfarin, and even fewer can claim an increase in use more than 50 years following introduction.

Warfarin is a Vitamin K antagonist. Gamma-carboxylation of vitamin K is crucial for coagulation factors II, VII, IX, and X to function properly, as well as antithrombotic endogenous Protein C and Protein S. Gamma-carboxylation of vitamin K allows these clotting proteins to bind calcium at phospholipid surfaces upon which coagulation occurs. Warfarin and other vitamin K antagonists interfere with vitamin K and cause the liver to synthesize nonfunctional coagulation factors.

Warfarin is almost completely absorbed by the gastrointestinal mucosa. It is metabolized in the liver by the Cytochrome P450 system. The kidney eliminates largely inactive metabolites.

Warfarin anticoagulation is prescribed to prevent stroke and venous thromboembolism. Optimal dosing requires achieving and maintaining a target range International Normalized Ratio (INR). The INR itself is a prothrombin time that is standardized according to the type of thromboplastin reagent used by the coagulation laboratory. Each thromboplastin reagent has a designated International Sensitivity Index. The formula used to calculate the INR is shown below:

The target INR for most indications, including atrial fibrillation, DVT, and pulmonary embolism, is usually between 2.0 and 3.0.

Excessive dosing is characterized by an elevated INR and precipitates hemorrhage, including stroke due to intracranial bleeding. To minimize the risk of intracranial hemorrhage, it is important to maintain a maximum INR level of 3.0. When the INR exceeds 3.0, the risk of intracranial bleeding increases exponentially.

Inadequate dosing, associated with a subtherapeutic INR, predisposes to stroke due to thromboembolism and to DVT or pulmonary embolism. For example, to prevent a thrombotic stroke in patients with atrial fibrillation, it is important to maintain an INR of at least 2.0.

The most vulnerable period for thrombosis and hemorrhage due to warfarin is during the initiation phase of anticoagulation, when optimal dosing is least certain. Adverse event rates are highest during this vulnerable period, which is generally considered to persist for at least 3 months. Patients who have not been previously exposed to warfarin are most vulnerable because there is no individual history to guide the clinician on an optimal initiation dose for those particular patients.

Dosing nomograms work poorly. Trial and error predominates as the method of dosing warfarin. Warfarin is virtually the only contemporary drug prescribed using trial and error methodology.

Various warfarin initiation regimens have been attempted, but none are in common use. In 1984, Fennerty proposed an every 16-hour dosing initiation nomogram for patients with venous thromboembolism whose average age was 52 years. This nomogram never gained wide support because of the awkward dosing interval and because it had been used in a patient population much younger than the average population of patients who take warfarin. In 1998, the "modified Fennerty" nomogram was introduced and dosed patients with warfarin every 24 hours. The nomogram enrolled an older population, average age of 78 years. However, 35% of these patients had excessively high INRs that exceeded 4.0 within the first 4 days of warfarin initiation.

Many clinical factors predispose to an excessively high INR: advanced age, abnormal liver function, decreased vitamin K intake because of poor nutrition or poor appetite, diarrhea, antibiotics, certain other concomitant medications, alcohol in binges, and perhaps changes in warfarin preparation (substituting one generic preparation for another or interchanging generic with brand-name Coumadin®). The most common reason for abnormally low INRs is intake of high amounts of vitamin K from green leafy vegetables, certain drug-warfarin interactions, or failure to take warfarin appropriately.

ADVANCES IN GENETICS:

Genotyping patients at the onset of warfarin anticoagulation may allow more precise dosing. This may translate into fewer major bleeding and clotting events as well as fewer out-of-target-range INRs, which serve as a surrogate for bleeding and clotting complications. During the first several weeks following prescription of warfarin, INR laboratory tests are obtained frequently, often twice weekly. Better predictive assessment of the optimal dose will decrease laboratory costs and improve convenience for patients.

Cytochrome P450 2C9 genotyping can identify mutations associated with impaired warfarin metabolism. The CYP2C9 genotype accounts for about 10% of warfarin dose variance. Vitamin K receptor polymorphism testing can identify whether patients require low, intermediate, or high doses of warfarin. Five common vitamin K receptor gene haplotypes account for about an additional 25% of warfarin dose variance.

Until now, the major drawback in applying screening for CYP2C9 polymorphisms to warfarin dosing and VKORC1 genotyping has been slow turnaround time. However, the HPCGG will be able in the Nomogram Development Trial to offer turnaround within 24-48 hours. This rapid turnaround time will allow initial immediate anticoagulation with once or twice daily injectable agents for several days. Therefore, prior to the initiation of warfarin, there will be sufficient time for the genetic information to be received and implemented by the clinical team.

The human cytochrome P450 (CYP) superfamily comprises 57 genes. These genes code for a myriad of enzymatic reactions. The cytochrome P450 CYP2C9 is responsible for metabolism of the S enantiomer of warfarin. Two allelic variants, CYP2C9*2 and CYP2C9*3, differ from the wild type CYP2C9*1 by a single amino acid substitution. The allelic variants are associated with impaired hydroxylation of S-warfarin.

A retrospective cohort study of 200 patients receiving warfarin dosed by anticoagulation clinics suggested that the CYP2C9*2 and CYP2C9*3 polymorphisms are associated with an increased risk of excessive anticoagulation and of bleeding events.

At the Brigham and Women's Hospital Anticoagulation Service, we identified 73 patients for CYP2C9 genotyping, which we assessed with PCR amplification and restriction enzyme digestion analysis of DNA isolated from circulating leukocytes. The CYP2C9 polymorphisms independently predicted low warfarin requirements after adjusting for body mass index, age, acetaminophen use, and race. At least one polymorphism was present in every patient requiring 1.5 mg or less of daily warfarin. We did find higher rates of excessive anticoagulation but did not observe higher bleeding rates in patients with these polymorphisms.

To date, only one prospective study has been published on warfarin dosing based upon cytochrome P450 2C9 genotyping. It was a negative study that failed to prove the hypothesis that genotyping would lead to better control of warfarin dosing. 48 orthopedic surgery patients were studied with genotyping and screening for nongenetic factors that might affect warfarin dosing and bleeding risk. The warfarin dosing algorithms based upon the genetic screening led to achievement of a stable and therapeutic INR in both the wild type group and the CYP2C9 variant groups with a similar time course. Nevertheless, despite pharmacogenetics-based dosing, patients with variants were at higher risk for excessive anticoagulation, defined as an INR greater than 4.0.

This failed study emphasizes the pivotal importance of a comprehensive nomogram development phase prior to initiating a randomized controlled trial. This trial also demonstrates the need to consider other factors that affect the INR and warfarin dose: advanced age, underlying comorbidities and thrombotic disposition, abnormal liver function, inadequate or excessive vitamin K intake, altered vitamin K metabolism (e.g., diarrhea or antibiotics), alcohol and drug-food interactions, and changes in warfarin preparation (switching among different generics or switching to or from brand name Coumadin®). The most important lesson from this cohort study is that to decrease clinical adverse events due to warfarin, it is first necessary to develop a warfarin nomogram that is superior than the current practice of educated guesses and trial and error.

Rieder and colleagues have identified 10 non-coding single- nucleotide polymorphisms (SNPs) in the vitamin K epoxide reductase complex 1 (VKORC1) gene that fall into five major haplotypes. Two of these haplotypes, A and B, can be used to determine whether patients require low (AA, 2.7 mg/day), intermediate (AB, 4.9 mg/day), or high (BB, 6.2 mg/day) doses of drug. The haplotypes differ according to racial distribution. These haplotypes are responsible for 25% of the variance in dose. Therefore, a combination of cytochrome P450 and VKORC1 genotyping will facilitate optimal warfarin dosing.

OBJECTIVE:

Primary Objective:

We will develop a nomogram for warfarin dosing that uses rapid turnaround genetic testing and monthly nomogram modification (if necessary) to achieve effective and safe warfarin induction and maintenance. More than 70% of the time, we will maintain warfarin naïve patients within the target therapeutic range. The percent of time in the therapeutic range will be analyzed beginning 2 weeks after initiation of warfarin. Analyses will be stratified by the indication for anticoagulation.

We will obtain Informed Consent for exploratory genetic testing of the sampled DNA, in addition to cytochrome P450 2C9 and VKORC1 alleles. This flexible approach will permit us to add additional promising tests that emerge and so that we can modify the nomogram to make it even more effective in achieving the target range for the INR.

PLANS:

Genetic Testing:

1. Detect known alleles of cytochrome P450 and Vitamin K epoxide reductase complex 1 (VKORC1).
2. Collect 5 ml of blood into EDTA (lavender top) tubes.
3. DNA will be processed using the ROCHE MagnaPure automated prep system.

Patient Population:

Warfarin naïve patients undergoing initiation of warfarin anticoagulation at participating Partners anticoagulation clinics, including Brigham and Women's Hospital, Massachusetts General Hospital, North Shore Medical Center, Faulkner Hospital, Spaulding Rehabilitation Hospital, and Newton Wellesley Hospital.

Overview and Timeline:

We will enroll patients over 9 months, follow each patient for 3 months with twice weekly coagulation testing of the prothrombin time standardized to the International Normalized Ratio, and adjust monthly the nomogram (if necessary) to improve the fit with emerging data from the cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Any newly diagnosed condition that will require treatment with therapeutic doses of warfarin for at least 4-6 weeks, e.g. deep venous thrombosis (DVT), pulmonary embolism (PE), atrial fibrillation (AF), orthopedic surgery, etc.
3. Written informed consent

Exclusion Criteria:

1. Current treatment with warfarin
2. Contraindication to therapeutic anticoagulation:

   * Active major bleeding
   * History of intracranial bleeding
   * Surgery, delivery, organ biopsy within 3 days
   * Gastrointestinal bleeding within 10 days
   * Major trauma within 3 days
   * Head injury requiring hospitalization within 3 months
   * Intracranial tumor
   * Neurosurgery or ophthalmologic surgery within the past month
3. Life expectancy < 3 months
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Creager, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Fennerty A, Dolben J, Thomas P, Backhouse G, Bentley DP, Campbell IA, Routledge PA. Flexible induction dose regimen for warfarin and prediction of maintenance dose. Br Med J (Clin Res Ed). 1984 Apr 28;288(6426):1268-70. doi: 10.1136/bmj.288.6426.1268. PMID 6424820
- [Background] Cooper MW, Hendra TJ. Prospective evaluation of a modified Fennerty regimen for anticoagulating elderly people. Age Ageing. 1998 Sep;27(5):655-6. doi: 10.1093/ageing/27.5.655. No abstract available. PMID 12675109
- [Background] Nebert DW, Russell DW. Clinical importance of the cytochromes P450. Lancet. 2002 Oct 12;360(9340):1155-62. doi: 10.1016/S0140-6736(02)11203-7. PMID 12387968
- [Background] Aithal GP, Day CP, Kesteven PJ, Daly AK. Association of polymorphisms in the cytochrome P450 CYP2C9 with warfarin dose requirement and risk of bleeding complications. Lancet. 1999 Feb 27;353(9154):717-9. doi: 10.1016/S0140-6736(98)04474-2. PMID 10073515
- [Background] Higashi MK, Veenstra DL, Kondo LM, Wittkowsky AK, Srinouanprachanh SL, Farin FM, Rettie AE. Association between CYP2C9 genetic variants and anticoagulation-related outcomes during warfarin therapy. JAMA. 2002 Apr 3;287(13):1690-8. doi: 10.1001/jama.287.13.1690. PMID 11926893
- [Background] Joffe HV, Goldhaber SZ. Effectiveness and safety of long-term anticoagulation of patients >/=90 years of age with atrial fibrillation. Am J Cardiol. 2002 Dec 15;90(12):1397-8. doi: 10.1016/s0002-9149(02)02883-7. No abstract available. PMID 12480055
- [Background] Fanikos J, Grasso-Correnti N, Shah R, Kucher N, Goldhaber SZ. Major bleeding complications in a specialized anticoagulation service. Am J Cardiol. 2005 Aug 15;96(4):595-8. doi: 10.1016/j.amjcard.2005.03.104. PMID 16098319
- [Background] Joffe HV, Xu R, Johnson FB, Longtine J, Kucher N, Goldhaber SZ. Warfarin dosing and cytochrome P450 2C9 polymorphisms. Thromb Haemost. 2004 Jun;91(6):1123-8. doi: 10.1160/TH04-02-0083. PMID 15175798
- [Background] Voora D, Eby C, Linder MW, Milligan PE, Bukaveckas BL, McLeod HL, Maloney W, Clohisy J, Burnett RS, Grosso L, Gatchel SK, Gage BF. Prospective dosing of warfarin based on cytochrome P-450 2C9 genotype. Thromb Haemost. 2005 Apr;93(4):700-5. doi: 10.1160/TH04-08-0542. PMID 15841315
- [Background] Rieder MJ, Reiner AP, Gage BF, Nickerson DA, Eby CS, McLeod HL, Blough DK, Thummel KE, Veenstra DL, Rettie AE. Effect of VKORC1 haplotypes on transcriptional regulation and warfarin dose. N Engl J Med. 2005 Jun 2;352(22):2285-93. doi: 10.1056/NEJMoa044503. PMID 15930419
- See also: North American Thrombosis Forum — http://www.natfonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Warfarin naïve patients undergoing initiation of warfarin anticoagulation at participating Partners anticoagulation clinics, including Brigham and Women's Hospital, Massachusetts General Hospital, North Shore Medical Center, Faulkner Hospital, Spaulding Rehabilitation Hospital, and Newton Wellesley Hospital.
Pre-assignment Details: We enrolled patients over 9 months, following each patient for 3 months with twice weekly coagulation testing of the prothrombin time standardized to the International Normalized Ratio, and adjusted monthly the nomogram (if necessary) to improve the fit with emerging data from the cohort.
Groups:
- Dosing Algorithm A: Algorithm A was a dosing decision-tree that included both clinical and genetic factors. It was based upon optimal clinical practice at the Brigham and Women's Hospital's Anticoagulation Management Service as well as published literature that has utilised warfarin pharmacogenetics.
  Doses were subsequently adjusted based on serial INR measurements.
- Dosing Algorithm B: Dosing Algorithm B was generated from an analysis of warfarin dose, INR, genetic factors, demographic factors and concomitant drug therapy from an initial prospective group of 74 patients treated using Algorithm A. Using these data, a mechanistic concentration-INR model was constructed to refine the estimates of the effect of CYP2C9 genotypes, VKORC1 haplotypes, age, and concomitant medications.
- Dosing Algorithm C: Dosing Algorithm C was generated as an update of dosing Algorithm B and was based upon additional patient data, similar to what was described above for Algorithm B, from the prospective accrual of 203 patients in the CROWN trial. The major difference between Algorithm B and Algorithm C was an update of the half maximal inhibitory concentration (IC50) estimate for each VKORC1 haplotype in the model used to generate Algorithm B to reflect warfarin's PD effect as evident in the acquired patient data. Simulations using Algorithm C were repeated using the clinical endpoints described above to derive the optimal starting warfarin doses and titration scheme that was tested prospectively in subsequent patients enrolled in the CROWN study.
Period: Overall Study
Arm/Group | Dosing Algorithm A | Dosing Algorithm B | Dosing Algorithm C
Started | 118 | 147 | 79
Completed | 118 | 147 | 79
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dosing Algorithm A: Three dosing algorithms (A, B, and C, respectively) were used in this investigation. The algorithms were developed sequentially to select both an initial warfarin dose and a titration scheme intended to maximise the likelihood of achieving and maintaining the target INR. The algorithms were refined using adaptive methods that allow for continual reassessment of patient-level data to optimize the predictive power of the algorithms. Algorithm A was a dosing decision-tree that included both clinical and genetic factors. It was based upon optimal clinical practice at the Brigham and Women's Hospital's Anticoagulation Management Service as well as published literature that has utilised warfarin pharmacogenetics.
  Doses were subsequently adjusted based on serial INR measurements.
- Dosing Algorithm B: Three dosing algorithms (A, B, and C, respectively) were used in this investigation. The algorithms were developed sequentially to select both an initial warfarin dose and a titration scheme intended to maximise the likelihood of achieving and maintaining the target INR. The algorithms were refined using adaptive methods that allow for continual reassessment of patient-level data to optimize the predictive power of the algorithms. Dosing Algorithm B was generated from an analysis of warfarin dose, INR, genetic factors, demographic factors and concomitant drug therapy from an initial prospective group of 74 patients treated using Algorithm A. Using these data, a mechanistic concentration-INR model was constructed to refine the estimates of the effect of CYP2C9 genotypes, VKORC1 haplotypes, age, and concomitant medications.
- Dosing Algorithm C: Three dosing algorithms (A, B, and C, respectively) were used in this investigation. The algorithms were developed sequentially to select both an initial warfarin dose and a titration scheme intended to maximise the likelihood of achieving and maintaining the target INR. The algorithms were refined using adaptive methods that allow for continual reassessment of patient-level data to optimize the predictive power of the algorithms. Dosing Algorithm C was generated as an update of dosing Algorithm B and was based upon additional patient data, similar to what was described above for Algorithm B, from the prospective accrual of 203 patients in the CROWN trial. The major difference between Algorithm B and Algorithm C was an update of the half maximal inhibitory concentration (IC50) estimate for each VKORC1 haplotype in the model used to generate Algorithm B to reflect warfarin's PD effect as evident in the acquired patient data.
- Total: Total of all reporting groups
Arm/Group | Dosing Algorithm A | Dosing Algorithm B | Dosing Algorithm C | Total
Number analyzed (Participants) | 118 | 147 | 79 | 344
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 118 | 147 | 79 | 344
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 64.7 (16.6) | 57.9 (16.5) | 57.2 (15.6) | 60.1 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 64 | 38 | 162
  Male | 58 | 83 | 41 | 182
Region of Enrollment [Number; unit: participants]
  United States | 118 | 147 | 79 | 344

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Time That INR Within Therapeutic Range Using Linear Interpolation (Rosendaal et al).
Description: Primary end point: mean percentage of time INR is within therapeutic range. Though target INR was 2.0-3.0, therapeutic INR is considered 1.8-3.2 (allows for INR measurement error and avoids problems inherent in overcorrection).
  The international normalized ratio (INR) is one way of presenting prothrombin time test results for people taking the blood-thinning medication warfarin. The INR formula adjusts for variation in laboratory testing methods so that test results can be comparable.
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Dosing Algorithm A | Dosing Algorithm B | Dosing Algorithm C
Number analyzed (Participants) | 118 | 147 | 79
percentage of time | 58.9 (22) | 59.7 (23) | 65.8 (16.9)

2. Secondary Outcome: Time to the First Therapeutic INR.
Description: The INR (international normalized ratio) is a derived measure of the prothrombin time. In this trial, a therapeutic INR was considered 1.8 to 3.2
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dosing Algorithm A | Dosing Algorithm B | Dosing Algorithm C
Number analyzed (Participants) | 118 | 147 | 79
Days | 9.1 (4.5) | 10.4 (4.9) | 9.7 (4.4)

3. Secondary Outcome: Per-patient Percentage of INRs Out of the Therapeutic Range
Description: as for outcome 2
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: percentage of INRs out of range
Arm/Group | Dosing Algorithm A | Dosing Algorithm B | Dosing Algorithm C
Number analyzed (Participants) | 118 | 147 | 79
percentage of INRs out of range | 42.2 (21.6) | 37.7 (22.8) | 33.3 (16.8)

4. Secondary Outcome: Time to Stable Anticoagulation (in Days).
Description: Defined as two consecutive INRs within the therapeutic range >7 days apart and with no dose change during this time.
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dosing Algorithm A | Dosing Algorithm B | Dosing Algorithm C
Number analyzed (Participants) | 118 | 147 | 79
Days | 50.8 (20.1) | 34.6 (14.9) | 31.5 (13.1)

5. Secondary Outcome: Proportion of Patients With Serious Adverse Clinical Events.
Description: Defined as an INR>4.0, use of vitamin K, major bleeding events (as defined by the Thrombolysis in Myocardial Infarction [TIMI] criteria), thromboembolic events, stroke (all cause), myocardial infarction, and death (all cause).
Time Frame: 90 Days
Measure: Number; unit: participants
Arm/Group | Dosing Algorithm A | Dosing Algorithm B | Dosing Algorithm C
Number analyzed (Participants) | 118 | 147 | 79
participants | 43 | 41 | 24

ADVERSE EVENTS:
Time Frame: 90 Days
Arm/Group | Dosing Algorithm A | Dosing Algorithm B | Dosing Algorithm C
Serious Adverse Events (participants affected / at risk) | 43/118 | 41/147 | 24/79
Other Adverse Events (participants affected / at risk) | 0/118 | 0/147 | 0/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dosing Algorithm A (N=118) | Dosing Algorithm B (N=147) | Dosing Algorithm C (N=79)
INR ≥ 4 (Vascular disorders) | 39 (39) | 36 (36) | 22 (22)
Major bleeding events (TIMI definition) (Vascular disorders) | 2 (2) | 3 (3) | 2 (2)
Vitamin K administration (Investigations) | 2 (2) | 0 (0) | 0 (0)
Thrombotic events (MI, stroke, VTE) (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No